CLINICAL TRIAL: NCT04427748
Title: The Change of Electrophysiology in Congenital Cataract After Lensectomy and Anterior Vitrectomy
Brief Title: Electrophysiology in Congenital Cataract After Lensectomy and Anterior
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Clinical professor, Wenzhou Medical University
Other Study IDs: Electrophysiology-WJJ
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Congenital Cataract
Keywords: ERG

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- congenital cataract group: children with congenital cataract who underwent lensectomy and anterior vitrectomy and IOL implantation are perfomed ERG
- age-matched normal children group: age-matched normal children are perfomed ERG

SUMMARY:
In this prospective study , a cohort of 91 eyes with congenital cataract and 25 eyes normal eyes from Wenzhou medical university was erolled.91 eyes with congenital cataract was after lensectomy and anterior vitrectomy as test group, 25 normal eyes as control group. The a- and b-wave and PhNR related parameters was evaluated.

DETAILED DESCRIPTION:
Secondary IOL implantation in aphika children and lensectomy and anterior vitrectomy and primary IOL implantation in children with congenital cataract were both performed by the same surgeon(Z.Y.E).

electroretinography and photopic negative response are performed to each patient.The research was to evaluate the relationship between the best corrected visionn and the related parameters of a- and b-wave and PhNR .

ELIGIBILITY:
Inclusion Criteria:

* phakic children diagnosed with congenital cataract who underwent secondary IOL implantation and children with congenital cataract who underwent lensectomy and anterior vitrectomy and primary IOL implantation

Exclusion Criteria:

* patients with mild cataracts do not require surgery

Ages: 18 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: congenital cataract age from 1.5 years to 15 years who underwent cataract surgery at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
ERG | at least 1year after the surgery of congenital cataract
  investigate retinal function changes of congenital cataract children. ERG related parameters including a- and b-wave and PhNR amplitude and latency.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hosptial of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Wang J, Wang Y, Guan W, Zhao YE. Full-field electroretinogram recorded with skin electrodes in 6- to 12-year-old children. Doc Ophthalmol. 2023 Dec;147(3):179-188. doi: 10.1007/s10633-023-09944-9. Epub 2023 Aug 2. PMID 37530953